CLINICAL TRIAL: NCT02665806
Title: Ciclesonide vs Fluticasone Propionate Nasal Sprays in Patients With Nasal Poplyposis; a Randomized Clinical Trial
Brief Title: Ciclesonide vs Fluticasone Nasal Sprays in Nasal Poplyposis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohsen Naraghi, Assistant Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.TUMS.REC.1394.1586
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Rhinosinustis With Polyps
Keywords: Ciclesonide; Fluticasone propionate; Nasal Polyposis; Chronic Sinuitis; Chronic rhinosinusitis
MeSH Terms: conditions — Nasal Polyps | interventions — ciclesonide; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ciclesonide (Experimental)
  Interventions: Drug: Ciclesonide
- Fluticasone (Active Comparator)
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Ciclesonide — intranasal ciclesonide spray 200 µg once daily
  Arms: Ciclesonide
Drug: Fluticasone — fluticasone propionate aqueous nasal spray 200 µg twice a day
  Arms: Fluticasone

SUMMARY:
This study is designed to compare ciclesonide nasal spray once daily with fluticasone propionate aquas nasal spray BD, which is commonly prescribed in patients with nasal polyposis, in order to relieve symptoms of these patients.

DETAILED DESCRIPTION:
The study will be conducted in a tertiary ENT center in Tehran. Endoscopic severity grades for patients will be determined for polyps on the basis of 3 point classification system: 1, confined to middle meatus; 2, below level of middle turbinate; 3, causing total obstruction. Also, patients will be undergone paranasal sinus CT scan to determine Lund-Mackay stage which defined by sum of scores of each of 12 paranasal sinuses (0 for a completely lucent, 1 for a partially opaque and 2 for a completely opaque sinus). Patients will be randomized to treat in one of two groups: 1 month of therapy with fluticasone propionate aqueous nasal spray (FPANS) 200 µg twice a day or 1 month of therapy with intranasal ciclesonide spray 200 µg once daily. All patients will be given written, easy to understand instruction about how to use nasal sprays. All included patients are asked to answer the disease specific Persian language validated SNOT20 quality of life questionnaire to evaluate symptom severity before starting the treatment. SNOT20 is a symptom severity and health related quality of life measure in sinonasal diseases that contains 20 questions about CRS related symptoms. Symptoms severity is scored 0, indicating no problem to 5, indicating worst possible symptom. Then scores of each of 20 items will be added to produce a total score ranging from 0 to 100. After one month of treatment patients will be visited by a blind physician to assess the symptoms. Then patients will answer the SNOT20 questionnaire again. Patients will be given a chance to report any problem during drug administration and enquired about adverse effects at the end of 1 month of treatment by the physician. Withdrawals is defined as any drug or study discontinuation due to adverse effects or lack of efficacy.

By considering 5% level of significance, to have 90% power to detect a clinically important difference of 0.6 points between two groups in improving total score of SNOT20 assuming a standard deviation (SD) of 0.6, we should include 22 cases in each study arm. To address a 10% probable loss to follow up, we would recruit 24 cases in each arm.

The continuous variables will be shown as mean ± SD. The categorical variables will be presented as frequency and percentage. The normality of measure outcome variables will be tested graphically as well as statistically with the Shapiro-Wilk test. In case of normal distribution we would use parametric t-test to compare the mean values between two groups. Otherwise we would use non-parametric Mann-Whitney test. Chi-squared or Fischer-exact tests will be used to compare categorical variables. All the statistical analyses will be conducted using IBM SPSS statistics for Windows, version 23.0, (Armonk, NY: IBM Corp.).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with the diagnosis of symptomatic nasal polyposis included.
* Objective confirmation of chronic rhinosinusitis with polyps was done by paranasal sinuses CT scan and Endoscopy.

Exclusion Criteria:

* Administration of systemic corticosteroids during last 3 months Administration of antihistamines, nasal steroids 15 days prior the including to the study.
* History of surgical treatment during last 3 month.
* History of septal deviation, severe epistaxis, cystic fibrosis, severe or non-controlled asthma, current purulent nasal infection, allergic rhinitis.
* Hypersensitivity or contraindication to steroids.
* Any positive history that was suspected to influence study parameters.
* NP requiring systemic corticosteroids or daily use of saline irrigations.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
SNOT20 score difference | 1 Month
  The change from the baseline in SNOT20 total score after the treatment period

SECONDARY OUTCOMES:
SNOT20 score difference in variuos endoscopic grades | 1 Month
  The change from the baseline in SNOT20 total score after the treatment period in patients with various endoscopic grades
SNOT20 score difference in variuos Lund-Mackay score | 1 Month
  The change from the baseline in SNOT20 total score after the treatment period in patients with various paranasanl sinus CT Scan's Lund-Mackay scores

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Naraghi, MD, Principal Investigator — Tehran University of Medical Sciences, Department of Otolaryngology-Head and Neck Surgery, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No